CLINICAL TRIAL: NCT05658432
Title: The Effect of Exercise Program Via Tele Rehabilitation on the Disease Symptoms and Cardiopulmonary Fitness Level in Patients With Fibromyalgia
Brief Title: Effects of Exercise Program Via Tele Rehabilitation on Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yeşim Kurtaiş Aytür, MD, Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2407
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; cardiopulmonary fitness; exercise; telehealth; telerehabilitation
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, parallel assignment, superiority, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group will perform an exercise program including aerobic, range of motion, stretching exercises on zoom sessions of 45 minutes each, under the supervision of the investigator, following a prerecorded exercise video. They will exercise thrice a week for 8 weeks, in groups of five.
  Interventions: Other: Exercise via telehealth
- Active control (Active Comparator): Control group will have access to the same exercise video and guided for the first session. They will be asked to do the exercises at home, exact the same duration and frequency of the experimental group but without supervision, for 8 weeks.
  Interventions: Other: Exercise unsupervised

INTERVENTIONS:
Other: Exercise via telehealth — Same as arm/group description
  Arms: Intervention
Other: Exercise unsupervised — Same as arm/group description
  Arms: Active control

SUMMARY:
The goal of this randomized controlled clinical trial is to investigate the effects of a telehealth exercise program on pain, symptoms, and cardiopulmonary fitness level of patients with fibromyalgia compared to a home exercise program. The main questions aims to answer:

* Is telehealth exercise program is superior to unsupervised home exercise program in and increasing cardiopulmonary fitness level?
* Is telehealth exercise program is superior to unsupervised home exercise program in controlling symptoms? Women participants with fibromyalgia randomized to an intervention or comparison group. Intervention group will exercise via telehealth system under supervision. Comparison group will exercise alone at home.

Researchers will compare the effects of supervised telehealth exercise program and home exercise on pain, symptoms, and cardiopulmonary fitness level of patients with fibromyalgia.

DETAILED DESCRIPTION:
This study is a randomized, parallel, superiority, controlled trial. Participants will be female patients with fibromyalgia who are admitted to Fibromyalgia Out-patient Clinic of Ankara University, Faculty of Medicine, Physical Medicine and Rehabillitation Department. Eligible patients will be randomized to be allocated to one of the two groups, experiment or control. Both groups will be informed about the possible positive effects of exercise. The experimental group will perform an exercise program including aerobic, range of motion, stretching exercises on zoom sessions of 45 minutes each, under the supervision of the investigator, following a prerecorded exercise video. They will exercise thrice a week for 8 weeks, in groups of five. Control group will have access to the same exercise video and guided for the first session. They will be asked to do the exercises at home, exact the same duration and frequency of the experimental group but without supervision, for 8 weeks. The control group will be called first once a week, than once in two weeks to remind exercising and fill out their exercise diary. All patients will be assessed by VAS for pain, Fibromyalgia Impact Questionnaire (FIQ), Hospital Anxiety and Depression Scale (HADS), cardiopulmonary exercise test and 6 min. walking test (6MWT) before and at the end of 8-weeks exercise program. Other symptoms related to fibromyalgia such as fatigue, sleep etc will also be recorded. Primary outcome measure is pain. Secondary outcome measures will be cardiopulmonary fitness level (VO2max), functional physical activity level (6MWT), symptom severity, disease impact (FIQ), psychological status (HADS) and subjective assessment of general well-being. The study's hypothesis suggest that improvement will be superior in the experimental group without any side effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as fibromyalgia according to the 2016 revision to the 2010/2011 fibromyalgia diagnostic criteria
* not attended in any exercise program in the last 3 months
* written consent to participate in the study regardless of the allocation group
* eligibility for digital literacy

Exclusion Criteria:

* pregnancy or breastfeeding patients
* absolute or relative contraindications for exercise including cardiopulmonary, uncontrolled systemic and/or musculoskeletal conditions
* psychiatric or cognitive disorder that may hamper assessments and treatment
* lack of internet access

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-17 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Changes in Pain | 0 week, 8 week
  Visual Analogue Scale (VAS) for pain will be used to measure the amplitude of patients' pain with fibromyalgia which is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. A straight horizontal line of 100 mm will be used, of which the ends are defined as the extreme limits of pain orientated from the left (worst) to the right (best). 20 mm decrease in VAS pain is considered to be an clinically important improvement.

SECONDARY OUTCOMES:
Impact of fibromyalgia on daily activities | 0 week, 8 week
  Fibromyalgia Impact Questionnaire (FIQ) is an instrument developed to assess the current health status of women with the fibromyalgia syndrome in clinical and research settings. Survey evaluates the severity of the condition on the individual's functional capacity and the quality of life. Each item is scored 0 to 10 and the total scores range from 0 to 100, where higher values indicate more disease impact. Scores are expressed as follows: from 0 to 38 mild effect, from 39 to 58 moderate effect, and from 59 to 100 severe impact. FIQ and validated in 1991 by Burckhardt et al., revised by Bennett RM, et al, in 2009. Revised FIQ was translated and adapted for the Turkish version in 2010 by Ediz, et al.
Symptoms related to psychological status | 0 week, 8 week
  Hospital Anxiety and Depression Scale (HADS) was originally developed by Zigmond and Snaith (1983) and is commonly used to determine the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Zigmond and Snaith created this outcome measure specifically to avoid reliance on aspects of these conditions that are also common somatic symptoms of illness, for example fatigue and insomnia or hypersomnia. So; it was created as a tool for the detection of anxiety and depression in people with physical health problems. Turkish validation and reliability study was done by Aydemir, et al (1997).
Physical activity level | 0 week, 8 week
  Physical activity will be assessed by VO2max which is the gold standard and will be directly measured by cardiopulmonary exercise testing (CPET). Before CPET dynamic lung function will be measured, and the exercise test will be performed by using Modified Bruce protocol on treadmill until the maximal exertion. During exercise testing ACSM's standards and guidelines (2021) will be followed. Standard CPET parameters such as oxygen consumption at anaerobic threshold, respiratory exchange ratio, respiratory quotient, and metabolic equivalent of task (MET) VO2-AT, RER, RQ, MET will also be recorded besides VO2max.
Functional physical capacity | 0 week, 8 week
  Functional capacity will be assessed by 6 minute walking test (6MWT) which was developed by the American Thoracic Society and it was officially introduced in 2002, coming along with a comprehensive guideline. It is a sub-maximal exercise test used to assess endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The test was initially designed to help in the assessment of patient with cardiopulmonary issues. Gradually, it was introduced in numerous other conditions. It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation. The validity and reliability of the test in fibromyalgia was shown by King, et al 1999, Pankoff, at al 2000.

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Kurtais Aytur, Prof., MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)